CLINICAL TRIAL: NCT01597726
Title: Cervical Priming Before Dilation & Evacuation: a Randomized Controlled Trial
Brief Title: Cervical Priming Before Dilation & Evacuation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ibis Reproductive Health (Other)
Collaborators: University of Cape Town (Other); Tygerberg Hospital (Unknown); Safe Abortion Action Fund of the International Planned Parenthood Federation (Unknown); Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32020
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Abortion, Induced
Keywords: Abortion, Induced; Laminaria; Misoprostol; Pregnancy Trimester, Second
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol (Active Comparator)
  Interventions: Drug: Misoprostol
- Laminaria (Experimental)
  Interventions: Device: Laminaria

INTERVENTIONS:
Drug: Misoprostol — Misoprostol 400 mcg administered buccally approximately 3-6 hours prior to D&E, repeated once 3 hours after the first dose if needed
  Arms: Misoprostol
Device: Laminaria — Laminaria tents inserted into the cervix 18 to 24 hours prior to D&E
  Arms: Laminaria

SUMMARY:
The purpose of this study is to compare the efficacy of buccal misoprostol cervical priming to laminaria priming among women undergoing D&E at 13-20 weeks gestation in the Western Cape Province, South Africa

DETAILED DESCRIPTION:
As misoprostol is increasingly being used for cervical preparation, concerns about its use and about the proportion of women expelling the fetus prior to the D&E and other side effects mean that rigorous data on possible advantages of osmotic dilators are needed. To address this gap in the literature, we propose to perform an RCT comparing two methods of cervical preparation prior to D&E:

1. Misoprostol 400 mcg administered buccally approximately 3-6 hours prior to D&E, repeated once 3 hours after the first dose (a modified version of the current protocol)
2. Laminaria tents inserted into the cervix 18 to 24 hours prior to D&E

ELIGIBILITY:
Inclusion Criteria:

* Woman seeking TOP between 13 and 20 weeks gestation as determined by ultrasound
* Age 18 or greater
* Willingness to participate in randomized study
* Fluency in English, Afrikaans or Xhosa
* Ability to give informed consent
* Staying within one hour travel time of Tygerberg Hospital for the night prior to the D&E
* Ability to be contacted by telephone

Exclusion Criteria:

* Active cervicitis
* Multiple gestation
* Fetal demise confirmed by ultrasound examination
* History of bleeding disorder or current anticoagulation therapy
* Allergy to misoprostol
* Currently breastfeeding and unwilling or unable to temporarily discard milk
* More than one prior cesarean delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Proportion of women with fetal expulsion prior to dilation and evacuation | Prior to D&E procedure

SECONDARY OUTCOMES:
Proportion of women requiring additional dilation (manual or pharmacologic) | At time of D&E procedure
Duration of dilation and evacuation procedure | End of D&E procedure
Frequency of major complications | Recorded at TOP visit and/or follow-up visit (target 7 days after procedure)
  Major complications to include:
  * Death
  * Admission to the ward after the procedure
  * Readmission after discharge
  * Abdominal surgical procedure
  * Suspected uterine perforation
  * Seizure
  * Hemorrhage requiring transfusion
  * Loss to follow-up after placement of laminaria
Frequency of Minor Complications | Recorded at TOP visit and/or follow-up visit (target 7 days after procedure)
  Minor complications to include:
  * Hemorrhage not requiring transfusion
  * Infection requiring outpatient treatment
  * Trauma to cervix or vagina
  * Transfer to another facility to complete the procedure
  * Need for repeat surgical evacuation of the uterus

CONTACTS AND LOCATIONS:
Overall Officials: Judy Kluge, MBChB, Principal Investigator — Tygerberg Hospital
Locations (1):
- Tygerberg Hospital, Cape Town, South Africa

REFERENCES:
- [Derived] Constant D, Kluge J, Harries J, Grossman D. An analysis of delays among women accessing second-trimester abortion in the public sector in South Africa. Contraception. 2019 Sep;100(3):209-213. doi: 10.1016/j.contraception.2019.04.009. Epub 2019 Apr 25. PMID 31029655
- [Derived] Grossman D, Constant D, Lince-Deroche N, Harries J, Kluge J. A randomized trial of misoprostol versus laminaria before dilation and evacuation in South Africa. Contraception. 2014 Sep;90(3):234-41. doi: 10.1016/j.contraception.2014.05.003. Epub 2014 May 14. PMID 24929888
- See also: Click here to visit the Ibis Reproductive Health website — http://www.ibisreproductivehealth.org/